CLINICAL TRIAL: NCT00005634
Title: Phase I Clinical and Pharmacological Study of Suberoylanilide Hydroxamic Acid- SAHA (MSK390) in Patients With Advanced Solid Tumors
Brief Title: Suberoylanilide Hydroxamic Acid in Treating Patients With Advanced Solid Tumors That Have Not Responded to Previous Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-059; CDR0000067789 (Registry Identifier: PDQ (Physician Data Query)); NCI-H00-0051
Record Dates: First submitted 2000-05-02; First posted 2003-12-17 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Prostate Cancer; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; small intestine lymphoma; recurrent prostate cancer; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; refractory hairy cell leukemia; chronic myelomonocytic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Prostatic Neoplasms; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — Vorinostat

INTERVENTIONS:
Drug: vorinostat

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of suberoylanilide hydroxamic acid in treating patients who have advanced primary or metastatic solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of suberoylanilide hydroxamic acid (SAHA) in patients with refractory malignancies. II. Assess the pharmacokinetic profile of SAHA in these patients. III. Assess the biologic effects of SAHA on normal tissues and on tumor cells in these patients.

OUTLINE: This is a dose-escalation study. Patients receive suberoylanilide hydroxamic acid (SAHA) IV over 2 hours on days 1-3. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity. Accelerated Phase: One patient per dose level receives escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which a patient experiences grade 2 or greater toxicity (other than hemoglobin anemia) with the first course or when 2 different patients experience a grade 2 toxicity (other than hemoglobin anemia) during any course of treatment. Standard Phase: Cohorts of 3-6 patients receive escalating doses of SAHA until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary or metastatic malignancy refractory to standard therapy or for which no curative therapy exists No progressive metastatic disease requiring palliative therapy within 4 weeks of study Progressive disease Increase in preexisting lesions on imaging or physical examination Patients with sole progression criterion of increased biochemical marker (e.g., carcinoembryonic antigen or CA 15-3) or increased symptoms not eligible Prostate cancer must be either progressive metastatic disease on imaging studies or have rising PSA values Minimum of 3 rising PSA values obtained at least 1 week apart, or 2 rising PSA values more than 1 month apart, with at least a 25% overall increase Serum testosterone less than 50 ng/mL Must maintain castrate status No active CNS or epidural tumor

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.0 mg/dL AST no greater than 37 U/L PT no greater than 14 seconds Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No significant cardiac disease No New York Heart Association class III or IV heart disease Pulmonary: No severe debilitating pulmonary disease Other: No infection requiring IV antibiotic treatment No other severe medical problems that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Recovered from prior biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered Endocrine therapy: Recovered from prior endocrine therapy Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy to target lesions Surgery: Not specified Other: At least 4 weeks since other prior investigational anticancer drugs and recovered No concurrent ketoconazole in patients with prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William K. Kelly, DO, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States